CLINICAL TRIAL: NCT06028828
Title: Risk-ADAPTed Conditioning Regimen for Allogeneic Hematopoietic Stem Cell Transplantation (ADAPT)
Brief Title: Risk-ADAPTed Conditioning Regimen for Allogeneic Hematopoietic Stem Cell Transplantation
Acronym: ADAPT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Stefan Octavian Ciurea, Professor of Clinical Medicine, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3095; UCI 21-90 (Other: UCI CFCCC)
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation; Allogeneic Stem Cell Transplantation; Hematologic Malignancies
Keywords: Allogeneic Hematopoietic Stem Cell Transplantation; Allogeneic Stem Cell transplantation; AHSCT; Hematologic malignancies; Melphalan; Hematopoietic stem cell transplant -composite risk
MeSH Terms: conditions — Hematologic Neoplasms | interventions — fludarabine; Melphalan; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with AML, ALL, MDS, CML, NHL, HD, CLL requiring AHSCT (Experimental): Patients will be treated with allogeneic stem cell transplantation (AHSCT) using fludarabine, melphalan and total body irradiation (TBI) conditioning with different melphalan and TBI doses based on their Hematopoietic Cell Transplant - Composite Risk (HCT-CR), age, and Karnofski performance status (KPS).
  Interventions: Drug: Fludarabine; Drug: Melphalan; Radiation: Total Body Irradiation

INTERVENTIONS:
Drug: Fludarabine — Given Day-5, Day-4, Day-3, Day-2
Drug: Melphalan — Given Day-5
Radiation: Total Body Irradiation — Given Day-1
  Other Names: TBI

SUMMARY:
This is a prospective, single-arm, phase II study. Patients will be treated with an allogeneic stem cell transplantation (AHSCT) using fludarabine, melphalan and total body irradiation (TBI) conditioning with different melphalan and TBI doses based on patient- and disease-related risk.

DETAILED DESCRIPTION:
Eligible patients will receive an allogeneic stem cell transplantation using a combination of fludarabine, melphalan and total body irradiation (TBI) conditioning regimen and post-transplant high dose cyclophosphamide (PTCY), tacrolimus and mycophenolate mofetil (MMF) for graft-versus-host prophylaxis.

Melphalan and TBI doses will be tailored based on the Hematopoietic Stem Cell Transplant- Composite Risk (HCT-CR), age and Karnofski performance status (KPS). Melphalan dose ranges from 100 -140 mg/m2 while TBI dose ranges from 2-5 Gy.

All patients will be monitored for safety and efficacy up to 2 years post-transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-70 years
2. Diagnosis of AML, ALL, MDS, CML, NHL, HD, CLL requiring AHSCT
3. Has an HLA-matched related (MRD), HLA-matched unrelated (MUD), haploidentical (HAPLO) or 1-Ag mismatched unrelated donor (MMUD)
4. Karnofsky performance >70%
5. Adequate major organ system function as demonstrated by:

   1. Serum creatinine clearance equal or more than 50 ml/min (calculated with Cockroft-Gault formula).
   2. Bilirubin equal or less than 1.5 mg/dl except for Gilbert's disease. ALT or AST equal or less than 200 IU/ml for adults. Conjugated (direct) bilirubin less than 2x upper limit of normal.
   3. Left ventricular ejection fraction equal or greater than 40%.
   4. Diffusing capacity for carbon monoxide (DLCO) equal or greater than 50% predicted corrected for hemoglobin.
6. Ability to understand and the willingness to sign a written informed consent. a. Both men and women and members of all races and ethnic groups are eligible for this trial. Non-English speaking, deaf, hard of hearing and illiterate individuals are eligible for this trial.

Exclusion Criteria:

1. Inability to comply with medical recommendations or follow-up
2. Pregnancy
3. Active/uncontrolled bacterial or viral infection (PI is the final arbiter of this criterion.)
4. Has active CNS or ocular disease involvement within 3 months
5. Patients with primary CNS lymphoma
6. Patients who require modifications of the conditional regimen

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 48 months
  PFS is defined as the time from stem cell infusion to time of disease relapse or death from any cause; data for patients who were alive without relapse will be censored at the date of last contact.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 48 months
  OS is defined as the time from stem cell infusion until death from any cause. Data of patients who were alive without relapse will be censored at the date of last contact.
Cumulative incidence of Graft-Versus-Host-Free, relapse-free survival (GRFS) | Up to 48 months
  GRFS is defined as time from stem cell infusion to time of the first event among acute GVHD grades 3-4, extensive chronic GVHD, relapse, and death. Data of patients who are event-free will be censored at the date of last contact.
Cumulative incidence of relapse | Up to 48 months
  Relapse is defined as re-occurrence of the disease after stem cell infusion. Cumulative incidence of relapse will be measured from date of stem cell infusion to date of disease relapse. Death without disease relapse is considered a competing risk for relapse. Data of patients who are alive without disease relapse will be censored at the date of last contact.
Cumulative incidence of Non-Relapse Mortality (NRM) | Up to 48 months
  NRM is defined as death related to AHSCT during continuous complete remission. Cumulative incidence of NRM will be measured from date of stem cell infusion to date of death. Disease relapse is considered a competing risk for NRM. Data of patients who are alive without disease relapse will be censored at the date of last contact.
Cumulative incidence of acute and chronic graft versus host disease (GVHD) | Up to 48 months
  Acute and chronic GVHD will be measured from date of stem cell infusion to date of the event. Death without GVHD is considered a competing risk for GVHD. Patients who are alive without GVHD will be censored at the date of last contact.
Area Under the Curve (AUC) of Melphalan | From melphalan infusion start time to 22 hours after the infusion.
  AUC will be used to determine the pharmacokinetic of melphalan after the infusion on D-5. Data will be summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan O. Ciurea, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, University of California Irvine, Orange, California, United States